CLINICAL TRIAL: NCT05557084
Title: Laparoscopic Clip-Gastroplasty With The Use Of Bariclip
Acronym: B-Clamp
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Gentileschi, Head of Department of Bariatric and Metabolic Surgery, University of Rome Tor Vergata
Other Study IDs: UNRome1
Record Dates: First submitted 2022-09-18; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Obesity, Abdominal; Surgery
Keywords: Bariclip; B-clamp; GERD; Bariatric Surgery; Obesity Surgery
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic vertical clip gastroplasty (LVCG) with Bariclip. — The investigator performed laparoscopic vertical clip gastroplasty, This procedure consists of a nonadjustable clip that is vertically placed around the stomach, parallel to the lesser curvature, mimicking the effect of sleeve gastrectomy. The clip restricts oral intake, the anatomy of the stomach is not permanently changed, the small bowel remains untouched, the digestive pathway is not diverted, no stapling or resection are required and the magnitude of restriction is supposed to remain constant during the years. The vertical clip is thus placed without risks of staple line leak, malabsorption side effects, changes in anatomy, and is potentially reversible [9]. creating a 4-cm window to enter the lesser sac while lifting the stomach to create sufficient space to be able to suture. Plication of the antrum for 3-5 cm is performed. Fluid testing for patency is performed with methylene blue or normal saline and the procedure is terminate.
  Other Names: Bariclip

SUMMARY:
Sleeve gastrectomy, the most commonly performed bariatric surgery procedure, carries limitations both short-term including postoperative complications such as hemorrhage and gastric fistula and long-term such as weight regain and gastro-esophageal reflux. A new procedure has been proposed to overcome many of these limitations: laparoscopic vertical clip gastroplasty (LVCG) with Bariclip. Primary outcome were major postoperative complications. Secondary outcomes included weight loss, incidence of de-novo GERD and comorbidity resolution.

DETAILED DESCRIPTION:
Methods. The investigators performed a review of data from a prospectively collected database. All patients submitted to primary LVCG were examined. Patients were submitted to LVCG Between July 2021 and March 2022. Collected data included demographic factors, pre-operative weight, pre-operative BMI, operative time, surgical complications, and clinical outcomes in terms of short and mid-term weight loss.

ELIGIBILITY:
Inclusion Criteria:

BMI > 40 BMI > 35 and comorbidities BMI > 30 with poorly controlled Diabetes mellitus II or hypertension

Exclusion Criteria:

Alcoholism Drug addiction Psychiatric Disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators performed a review of data from a prospectively collected database. All patients submitted to primary LVCG were examined. Patients were submitted to LVCG Between July 2021 and March 2022. Collected data included demographic factors, pre-operative weight, pre-operative BMI, operative time, surgical complications, and clinical outcomes in terms of short and mid-term weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
% Excess Weight Loss | 1 year
  Weight loss after laparoscopic vertical clip gastroplasty during the follow-up

SECONDARY OUTCOMES:
Post-operative complications | 1 year
  Complications occurred after laparoscopic vertical clip gastroplasty during the follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Michela Campanelli, Rome, RM
  - Department of Bariatric and Metabolic Surgery, San Carlo of Nancy Hospital and University of Rome "Tor Vergata", Rome, Italy, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noel P, Eddbali I, Nedelcu M. Laparoscopic Clip Gastroplasty with the BariClip. Obes Surg. 2020 Dec;30(12):5182-5183. doi: 10.1007/s11695-020-04803-x. PMID 32996101
- [Background] Noel P, Nedelcu AM, Eddbali I, Zundel N. Laparoscopic vertical clip gastroplasty - quality of life. Surg Obes Relat Dis. 2018 Oct;14(10):1587-1593. doi: 10.1016/j.soard.2018.07.013. Epub 2018 Jul 20. PMID 30449515